CLINICAL TRIAL: NCT00562172
Title: Lantus vs Sulfonylurea as add-on Therapy in Type 2 Diabetic Patients Failing Metformin Monotherapy: Comparison of Effects on Beta Cell Function and Metabolic Profile.
Brief Title: Insulin Glargine (Lantus) vs Sulfonylurea (SU) for BETA Cell Function (BETA Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_02193
Record Dates: First submitted 2007-11-15; First posted 2007-11-21 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Insulin glargine; Drug: Metformin
- 2 (Active Comparator)
  Interventions: Drug: Glimepiride; Drug: Metformin

INTERVENTIONS:
Drug: Insulin glargine — Once daily in the morning
  Arms: 1
Drug: Glimepiride — Once daily in the morning
  Arms: 2
Drug: Metformin — At least 1000 mg/day

SUMMARY:
Primary objective:

To compare long-term glycemic control and preservation of beta cell function when basal insulin or sulfonylurea is added on metformin in the early Type 2 Diabetes Mellitus patients

Secondary objective:

To assess the change of insulin resistance, microvascular complication incidence, patient satisfaction with treatment

ELIGIBILITY:
List of Inclusion and Exclusion Criteria:

Inclusion Criteria:

* Type 2 Diabetes Mellitus patients on metformin monotherapy
* 7% ≤ HbA1c ≤ 12%
* 20 kg/m² ≤BMI ≤ 35 kg/m²
* Diabetes duration: at least 6 months

Exclusion Criteria:

* Type 1 Diabetes Mellitus patients
* Clinical evidence of active liver disease, or serum Alanine AminoTransferase 3 times the upper limit of the normal range
* Serum creatinine: 1.5 mg/dl for males, 1.4 mg/dl for females
* Acute and chronic metabolic acidosis, including diabetic ketoacidosis
* History of alcohol or other substance abuse
* Pregnancy or not using contraceptive in childbearing aged women
* Known hypersensitivity to Lantus, SU or metformin
* Any disease or condition that in the opinion of the investigator may interfere with completion of the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
ß-cell Function parameter | From the signature of the Informed Consent Form (ICF) up to the end of study
Glucose Homeostasis and glycemic control status | From the signature of the Informed Consent Form (ICF) up to the end of study

SECONDARY OUTCOMES:
Insulin resistance parameter, Hypoglycemic episode, symptomatic, Weight change, Lipid profile, Inflammatory markers (CRP, Adiponectin, etcs), Patient satisfaction with diabetes treatment, Urine analysis, Creatinine | End of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Ahn, Study Director — Sanofi
Locations (1):
- Sanofi-aventis, Seoul, South Korea

REFERENCES:
- [Derived] Moon JS, Ha KS, Yoon JS, Lee HW, Lee HC, Won KC; BETA study group. The effect of glargine versus glimepiride on pancreatic beta-cell function in patients with type 2 diabetes uncontrolled on metformin monotherapy: open-label, randomized, controlled study. Acta Diabetol. 2014 Apr;51(2):277-85. doi: 10.1007/s00592-013-0553-z. Epub 2014 Jan 21. PMID 24445656